CLINICAL TRIAL: NCT02362308
Title: Glucose Metabolism in Subjects With Aldosterone-Producing Adenomas
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Collaborators: Brigham and Women's Hospital (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, James Matt Luther, James M Luther MD, MSCI, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Other Study IDs: 141553; R01DK096994 (NIH)
Record Dates: First submitted 2015-02-05; First posted 2015-02-12 (Estimated); Last update posted 2021-05-04 (Actual); Status verified 2021-04

CONDITIONS: Primary Aldosteronism
MeSH Terms: conditions — Hyperaldosteronism | interventions — Adrenalectomy; Mineralocorticoid Receptor Antagonists; Spironolactone; Eplerenone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Adrenalectomy: Subjects will undergo assessment before and after adrenalectomy for treatment of primary aldosteronism
  Interventions: Other: Adrenalectomy
- Medical Therapy: Subjects will undergo assessment before and after medical treatment of primary aldosteronism
  Interventions: Drug: mineralocorticoid receptor antagonist

INTERVENTIONS:
Other: Adrenalectomy — Adrenalectomy for treatment of primary aldosteronism, according to standard of care
  Groups: Adrenalectomy
Drug: mineralocorticoid receptor antagonist — Subjects will be treated with a mineralocorticoid receptor antagonist according to standard of care
  Other Names: spironolactone; eplerenone
  Groups: Medical Therapy

SUMMARY:
This observational study tests the hypothesis that endogenous aldosterone impairs insulin secretion and insulin sensitivity in subjects with primary aldosteronism.

DETAILED DESCRIPTION:
The week of each study period, subjects will be provided a standard 160mmol/d sodium diet for 6-8 days to control for inter-individual sodium intake.

In period 1, subjects will report after 5 days of controlled sodium diet for a hyperglycemic clamp study (to measure insulin secretion). Subjects will continue the study diet, and then return for a hyperinsulinemic-euglycemic clamp study (to measure insulin sensitivity).

After completion of period 1 assessment, subjects will undergo adrenalectomy by our endocrine surgeons or initiate medical treatment, according to routine clinical care.

In period 2, the investigators will repeat the studies in the same manner as period 1, 3 to 12 months after adrenalectomy or initiation of medical treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Ambulatory subjects, 18 to 70 years of age, inclusive
2. For female subjects, the following conditions must be met:

   * postmenopausal status for at least 1 year, or
   * status-post surgical sterilization, or
   * if of childbearing potential, utilization of adequate birth control and willingness to undergo urine beta-hcg testing on every study day.
3. Primary aldosteronism determined by both:

   * Biochemical hyperaldosteronism defined as either:

     1. Plasma aldosterone ≥15 ng/dL
     2. or aldosterone-to-renin ratio of ≥30 if on ACE inhibitor
     3. or aldosterone-to-renin ratio of ≥40 in absence of an ACE inhibitor
   * Positive suppression test defined as either:

     1. failure to suppress aldosterone to <7ng/dL after intravenous 0.9% saline infusion over 2 hours
     2. failure to suppress 24-hour urinary aldosterone excretion to <12 µcg with simultaneously documented urine sodium excretion >200 mmol.

Exclusion Criteria:

- Subjects presenting with any of the following will not be included in the study:

1. Previously diagnosed type 1 Diabetes
2. Type II Diabetes, as defined by ADA criteria:

   * Hemoglobin A1C ≥6.5%
   * Fasting plasma glucose ≥126mg/dl (7.0mmol/l)
   * 2-hour 75g oral glucose tolerance test (OGTT) plasma glucose ≥200mg/dl (11.1 mmol/l) d. Current treatment with anti-diabetic medication(s)
3. Impaired renal function [estimated glomerular filtration rate (eGFR) of <30ml/min] as determined by the four-variable Modification of Diet in Renal Disease (MDRD) equation, where serum creatinine (Scr) is expressed in mg/dl and age in years.
4. Prior allergies to medications used in the study protocol (e.g. L-arginine, potassium chloride, insulin), or to drugs within the same class.
5. Screening plasma potassium >5.5 mmol/L or sodium <135 mmol/L
6. Cardiovascular disease such as recent (<6 months) myocardial infarction, presence of angina pectoris, significant arrhythmia, congestive heart failure (LV hypertrophy acceptable), deep vein thrombosis, pulmonary embolism, second or third degree heart block, mitral valve stenosis, aortic stenosis or hypertrophic cardiomyopathy
7. Breast-feeding
8. Treatment with anticoagulants
9. History of serious neurologic disease such as cerebral hemorrhage, stroke, seizure, or transient ischemic attack
10. History or presence of immunological or hematological disorders
11. Diagnosis of asthma requiring use of inhaled beta agonist >1 time per week
12. Clinically significant gastrointestinal impairment that could interfere with drug absorption
13. Impaired hepatic function [aspartate amino transaminase (AST) and/or alanine amino transaminase (ALT) >2.0 x upper limit of normal range]
14. Hematocrit <35%
15. Any underlying or acute disease requiring regular medication which could possibly pose a threat to the subject or make implementation of the protocol or interpretation of the study results difficult, such as arthritis treated with non-steroidal antiinflammatory drugs
16. Treatment with chronic systemic glucocorticoid therapy (more than 7 consecutive days in 1 month)
17. Treatment with lithium salts
18. History of alcohol or drug abuse
19. Treatment with any investigational drug in the 1 month preceding the study
20. Mental conditions rendering the subject unable to understand the nature, scope and possible consequences of the study
21. Inability to comply with the protocol, e.g., uncooperative attitude, inability to return for follow-up visits, and unlikelihood of completing the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Change in Acute Glucose-stimulated Insulin Secretion | Change from Baseline vs. 3-12 months after intervention
  measured by hyperglycemic clamp
Change in Insulin Sensitivity Index | Change from Baseline vs. 3-12 months after intervention
  measured by hyperinsulinemic-euglycemic clamp
Change in Disposition Index (product of Insulin sensitivity index and acute insulin secretion) | Change from Baseline vs. 3-12 months after intervention
  Product of insulin sensitivity and insulin secretion

SECONDARY OUTCOMES:
Suppression of Hepatic glucose production | Change from Baseline vs. 3-12 months after intervention
  suppression of hepatic glucose production during hyperinsulinemic clamp, determined using glucose tracer

OTHER OUTCOMES:
Urinary exosomal biomarkers | Change from Baseline vs. 3-12 months after intervention
  Urinary biomarkers of renal sodium channels and sodium transporters
Associative learning Memory testing | Change from Baseline vs. 3-12 months after intervention
  Associative learning task matching images and words

CONTACTS AND LOCATIONS:
Overall Officials: James M Luther, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Result] Luther JM, Wei DS, Ghoshal K, Peng D, Adler GK, Turcu AF, Nian H, Yu C, Solorzano CC, Pozzi A, Brown NJ. Treatment of Primary Aldosteronism Increases Plasma Epoxyeicosatrienoic Acids. Hypertension. 2021 Apr;77(4):1323-1331. doi: 10.1161/HYPERTENSIONAHA.120.14808. Epub 2021 Feb 15. PMID 33583202
- [Result] Adler GK, Murray GR, Turcu AF, Nian H, Yu C, Solorzano CC, Manning R, Peng D, Luther JM. Primary Aldosteronism Decreases Insulin Secretion and Increases Insulin Clearance in Humans. Hypertension. 2020 May;75(5):1251-1259. doi: 10.1161/HYPERTENSIONAHA.119.13922. Epub 2020 Mar 16. PMID 32172621